CLINICAL TRIAL: NCT04722315
Title: Pilot Clinical Trial of Modified Atkins Diet for Kabuki Syndrome
Brief Title: Study of Modified Atkins Diet in Kabuki Syndrome
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00250195
Record Dates: First submitted 2020-11-24; First posted 2021-01-25 (Actual); Results first posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-04

CONDITIONS: Kabuki Syndrome
MeSH Terms: conditions — Kabuki syndrome

STUDY DESIGN:
Intervention Model Description: 15 participants with Kabuki syndrome will receive a 12 week dietary intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MAD diet group (Experimental): 15 adult participants with confirmed KMT2D pathogenic mutations. Baseline labs and education about Modified Atkins Diet. Then 12 weeks on a Modified Atkins Diet. Weekly urine dips for ketones and diet logs. Blood draw every 3 weeks.
  Interventions: Dietary Supplement: Modified Atkins diet

INTERVENTIONS:
Dietary Supplement: Modified Atkins diet — 12 weeks of modified Atkins diet

SUMMARY:
Animal models of Kabuki syndrome have showed a reversal of the cognitive phenotype with ketogenic diet. Modified Atkins diet is safer and easier tolerated than full ketogenic diet and still has the histone deacetylase inhibition believed to be responsible for the cognitive improvement. This study aims to examine a small number of adults with Kabuki syndrome before and after 12 weeks on a modified Atkins diet to determine if there is any cognitive improvement and if the diet can be tolerated.

DETAILED DESCRIPTION:
Consented participants will participate in an initial 2 day study visit. These participants will undergo cognitive and neurobehavioral testing and also will have baseline labs drawn and will meet with a Johns Hopkins nutritionist trained in modified Atkins diet for education. The labs are standard of care for diet initiation to rule out contraindications to the diet. Participants and/or their caregivers will keep a daily diet log and will be asked to download the free Carb Manager application onto their smartphone. They will send the logs and data back weekly. Participants will be given urine ketone strips and asked to use and record in their diet log twice weekly. Participants will have blood and urine samples collected locally every 3 weeks and sent back to study team to measure Beta-hydroxybutyrate, metabolic studies and methylation. Participants will return to Baltimore at the end of 12 weeks for a one day visit to repeat the cognitive assessment protocol, neurobehavioral measures, and repeat the initial and follow up lab tests.

ELIGIBILITY:
Inclusion Criteria:We will recruit 15 total participants with clinically-definite and genetically-confirmed Kabuki syndrome type 1 age 18 years and older. . will also be required.

* Clinical diagnosis of KS will be made based on recently published consensus diagnosis criteria
* Genetic confirmation of a pathogenic mutation in KMT2D

Exclusion Criteria:

* presence of another known genetic syndrome
* a health problem that would make a modified Atkins diet harmful
* inability to travel to Baltimore for 2 visits separated by 12 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2024-01-26 (Actual); Study Completion 2025-03-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Kennedy Krieger Institute, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- MAD Diet Group: 10 adult participants with confirmed KMT2D pathogenic mutations. Baseline labs and education about Modified Atkins Diet. Then 12 weeks on a Modified Atkins Diet.
  Modified Atkins diet: 12 weeks of modified Atkins diet
Period: Overall Study
Arm/Group | MAD Diet Group
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | MAD Diet Group
Number analyzed (Participants) | 10
Age, Continuous [Mean (Full Range); unit: years] | 24.9 [18 to 36]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Benton Judgement of Line Orientation
Description: Established measure to determine visuospatial perception. There are 30 items and each item is worth 1 point. Will assess change in score from baseline to post-diet. A higher score indicates a better performance (range 0-30).
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Baseline Measures: Baseline assessment of 10 adults with KMT2D pathogenic variants
- Measures After 12 Weeks of MAD: Assessment of 10 adults with KMT2D pathogenic variants after 12 weeks on Modified Atkins Diet
Arm/Group | Baseline Measures | Measures After 12 Weeks of MAD
Number analyzed (Participants) | 10 | 10
score on a scale | 8.6 (7.65) | 11.6 (8.11)

2. Primary Outcome: Brief Visuospatial Memory Test
Description: Established measure to determine visuospatial memory. Immediate scores range from 0 to 36 and a higher score indicates more correct responses. Delayed scores range from 0 to 12 and a higher score indicates more correct responses. Will assess change in score from baseline to post-diet.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Baseline BVMT Immediate Score: Total score of 3 immediate recall trials of BVMT
- Baseline BVMT Delayed Score: Total score of one delayed recall trial of BVMT
- BVMT Immediate Score Post-MAD: Total score of 3 immediate recall trials of BVMT after 12 weeks of MAD
- BVMT Delayed Score Post-MAD: Total score of one delayed recall trial of BVMT after 12 weeks of MAD
Arm/Group | Baseline BVMT Immediate Score | Baseline BVMT Delayed Score | BVMT Immediate Score Post-MAD | BVMT Delayed Score Post-MAD
Number analyzed (Participants) | 10 | 10 | 10 | 10
score on a scale | 10.9 (8.17) | 11.7 (8.29) | 4.1 (3.70) | 5 (3.83)

3. Primary Outcome: NIH Toolbox Picture Sequence Memory
Description: Established measure to determine visuospatial memory. Scaled scores based on age have a mean of 100 and a standard deviation of 15 and higher scores indicate more correct responses. Will assess change in this score from baseline to post-diet.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Baseline Measures | Measures After 12 Weeks of MAD
Number analyzed (Participants) | 10 | 10
score on a scale | 92.4 (14.23) | 93.2 (17.34)

4. Primary Outcome: Beery Developmental Test of Visual Motor Integration
Description: Established measure to determine visuomotor integration. Since these were all adults, raw scores were used. Range is 1-27. Higher scores indicate more correct responses. Will assess change in this score from baseline to post-diet.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: raw score
Arm/Group | Baseline Measures | Measures After 12 Weeks of MAD
Number analyzed (Participants) | 10 | 10
raw score | 16.3 (4.76) | 17.2 (4.16)

5. Primary Outcome: Beery Developmental Test of Visual Perception
Description: Established measure to determine visual perception. Since these were all adults, raw scores were used. Range is 1-27. Higher scores indicate more correct responses. Will assess change in this score from baseline to post-diet.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: raw score
Arm/Group | Baseline Measures | Measures After 12 Weeks of MAD
Number analyzed (Participants) | 10 | 10
raw score | 20.7 (3.02) | 21.2 (3.12)

6. Primary Outcome: Wechsler Intelligence Scale for Children -V Block Design
Description: Established measure to determine visuospatial processing. Since these were all adults, raw scores were used. Range is 0-66. Higher scores indicate more correct responses. Will assess change in this score from baseline to post-diet. Will assess change in this score from baseline to post-diet.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: raw score
Arm/Group | Baseline Measures | Measures After 12 Weeks of MAD
Number analyzed (Participants) | 10 | 10
raw score | 19.3 (8.37) | 21.4 (10.11)

7. Primary Outcome: Hopkins Verbal Learning Test
Description: Established measure to determine verbal memory. Scores range from 0 to 36 and a higher score indicates more correct responses. Will assess change in score from baseline to post-diet.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Baseline Measures | Measures After 12 Weeks of MAD
Number analyzed (Participants) | 10 | 10
score on a scale | 22.9 (6.98) | 24.3 (7.01)

8. Secondary Outcome: DNA Methylation Analysis
Description: Measure genome-wide methylation signature in blood of participants. To obtain genome-scale methylation measurements, bisulfite treated DNA from patient blood samples will be processed on the Infinium HumanMethylation450 BeadChip at the Johns Hopkins SNP Center in accordance with the manufacturer's recommendation. The Infinium HumanMethylation450 BeadChip measures DNA methylation levels at 485,512 loci across the genome. The array data will then be analyzed to get the proportion of methylation at a given CpG site from 0 to 1. These will be logit transformed to create M-values. Kabuki syndrome is known to have a unique signature methylation profile (determined by M-values across loci) that can be detected in blood. This genome wide DNA methylation will be done every 3 weeks to determine whether this signature changes with dietary therapy.
Time Frame: Every 3 weeks for 12 weeks
Reporting Status: Not Posted, anticipated posting 2025-07

9. Secondary Outcome: Caregiver Behavior Rating Scales: GAS-ID
Description: Rating scale for anxiety consists of 27 items with scores ranging from 0-70 with higher scores indicating more anxiety. Performed at baseline and post-diet.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Baseline Measures | Measures After 12 Weeks of MAD
Number analyzed (Participants) | 10 | 10
score on a scale | 12 (6.91) | 11.3 (6.27)

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Weekly calls to participants and labs (CBC, CMP, UA) at baseline and 12 weeks
Arm/Group | MAD Diet Group
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 7/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MAD Diet Group (N=10)
Diarrhea (Gastrointestinal disorders) | 3
Lightheadedness (General disorders) | 2
Hypertriglyceridemia or Hypercholesterolemia (Vascular disorders) | 3
Low platelets (Blood and lymphatic system disorders) | 2
Hypoglycemia (Endocrine disorders) | 1
Constipation (Gastrointestinal disorders) | 3

LIMITATIONS AND CAVEATS:
Single arm pilot study with no control group

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-01-31): https://cdn.clinicaltrials.gov/large-docs/15/NCT04722315/Prot_SAP_001.pdf
  • Informed Consent Form (2022-03-29): https://cdn.clinicaltrials.gov/large-docs/15/NCT04722315/ICF_000.pdf